CLINICAL TRIAL: NCT03891615
Title: Phase 1 Study of Niraparib in Combination With Osimertinib in EGFR-Mutated Advanced Lung Cancer
Brief Title: Niraparib in Combination With Osimertinib in EGFR-Mutated Advanced Lung Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Tesaro, Inc. (Industry)
Responsible Party: Principal Investigator, Zofia Piotrowska, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-613
Record Dates: First submitted 2019-03-25; First posted 2019-03-27 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Lung Cancer
Keywords: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — niraparib; osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Niraparib + Osimertinib (Experimental): * Niraparib will be administered orally once daily
  * Osimertinib will be administered by mouth once daily
  Interventions: Drug: Niraparib; Drug: Osimertinib

INTERVENTIONS:
Drug: Niraparib — Niraparib is a type of drug called a "PARP inhibitor", which blocks DNA (the genetic material of cells) damage from being repaired or may prevent damage from occurring in the first place. In cancer treatment, inhibiting PARP may help kill cancer cells through deadly DNA damage.
  Other Names: ZEJULA
Drug: Osimertinib — Osimertinib blocks mutated EGFR, which may cause tumor regression (when the tumor starts to shrink) and prevent the spread of the cancer.
  Other Names: Tagrisso

SUMMARY:
This research study is studying a combination of drugs as a possible treatment for EGFR-Mutated Advanced Lung Cancer.

The names of the study drugs involved in this study are Niraparib and Osimertinib.

DETAILED DESCRIPTION:
This research study is a Phase I clinical trial, which tests the safety of an investigational drug and also tries to define the appropriate dose of the investigational drug to use for further studies. "Investigational" means that the drug is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved niraparib for this specific disease but it has been approved for other uses.

The FDA has approved osimertinib as a treatment option for this disease.

Niraparib is a type of drug called a "PARP inhibitor", which blocks DNA (the genetic material of cells) damage from being repaired or may prevent damage from occurring in the first place. In cancer treatment, inhibiting PARP may help kill cancer cells through deadly DNA damage. PARP inhibition may be a treatment option for participants with this type of cancer due to altered repair and protection of tumor DNA.

Osimertinib is an inhibitor of the epidermal growth factor receptor (EGFR). In this type of cancer there is a mutation in the EGFR which is allowing the cancer to grow when it is not supposed to. Osimertinib blocks mutated EGFR, which may cause tumor regression (when the tumor starts to shrink) and prevent the spread of the cancer.

In this research study, the investigators are looking to see whether the combination of niraparib and osimertinib is safe and well tolerated and what the best dose of niraparib is in participants with EGFR-Mutated Advanced Lung Cancer. The investigators also hope that the combination of niraparib and osimertinib will stop the cancer from growing and spreading.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed stage IV (AJCC 8th ed.) NSCLC with an activating EGFR mutation as identified in a CLIA-approved laboratory.
* Presence of evaluable disease, either measure or non-measurable, in accordance with RECIST 1.1 criteria.
* Participants must have had clinical progression on osimertinib at any prior time, i.e., intervening therapy between osimertinib and study enrollment is allowed.
* Participants must have access to commercial osimertinib.
* Participants must not have received any prior PARP inhibitor therapy.
* Age minimum 18 years.
* ECOG performance status ≤1 (Karnofsky ≥70%, see Appendix A).
* Life expectancy of greater than 6 months.
* Participants must have normal organ and marrow function as defined below:

  * absolute neutrophil count ≥1,500/mcL
  * platelets ≥100,000/mcL
  * hemoglobin ≥ 9 g/dL
  * bilirubin total bilirubin ≤ 1.5 x upper limit of normal (ULN) (≤2.0 in patients with known Gilberts syndrome or liver metastases) OR direct bilirubin ≤ 1 x ULN
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal, unless liver metastases are present, in which case they must be ≤ 5 x ULN
  * creatinine ≤ 1.5 x institutional ULN OR
  * creatinine clearance ≥50 mL/min using the Cockcroft-Gault equation
* Participants must have undergone a prior tumor biopsy upon clinical progression on osimertinib. If it was not feasible or medically safe to undergo a biopsy a patient may enroll with permission of the PI.
* The effects of Niraparib on the developing human fetus are unknown but based on its mechanism of action Niraparib may cause fetal harm when administered to a pregnant woman. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry through 180 days after the last dose of study treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of Niraparib administration.
* Female participant must have a negative urine or serum pregnancy test within 7 days prior to taking study treatment if of childbearing potential, or is of nonchildbearing potential. Nonchildbearing potential is defined as follows (by other than medical reasons):

  --≥ 45 years of age and has not had menses for >1 year
  * Patients who have been amenorrhoeic for <2 years without history of a hysterectomy and oophorectomy must have a follicle stimulating hormone value in the postmenopausal range upon screening evaluation
  * Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure, otherwise the patient must be willing to use 2 adequate barrier methods throughout the study, starting with the screening visit through 180 days after the last dose of study treatment. See Section 4.4 for a list of acceptable birth control methods. Information must be captured appropriately within the site's source documents. Note: Abstinence is acceptable if this is the established and preferred contraception for the patient.
* Ability to take oral medications whole.
* Participant receiving corticosteroids may continue as long as their dose is stable for least 4 weeks prior to initiating protocol therapy.
* Participant must agree to not donate blood during the study or for 90 days after the last dose of study treatment
* Participant must agree not to breastfeed during the study or for 180 days after the last dose of study treatment.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants must not be simultaneously enrolled in any interventional clinical trial.
* Participants receiving any systemic standard of care or investigational therapy within 4 weeks from the last dose prior to planned study treatment, with the exception of osimertinib. This time frame may be shortened for participants depending on the characteristics of the individual therapy, after discussion with the Study PI. For investigational therapy, the time frame will not be shortened to less than at least 5 half-lives of the investigational agent.
* Patients receiving radiation therapy encompassing > 20% of the bone marrow by investigator's estimate within 14 days, or any radiation therapy within 7 days from the last treatment prior to planned study treatment. However, small volume palliative radiation therapy with no or little bone marrow exposure is allowed at the investigator's discretion.
* Participants may receive a stable dose of bisphosphonates for bone metastases, before and during the study as long as these were started at least 4 weeks prior to treatment.
* Participants who had any major surgery within the past 3 weeks (excluding vascular access placement, mediastinoscopy, or biopsies performed by an interventional service) and participant must have recovered from any surgical effects.
* Participants with symptomatic uncontrolled brain or leptomeningeal metastases. Participants with brain metastases that have been treated with prior radiation therapy and are stable on a subsequent scan are allowed. Participants with untreated possible brain metastases that are ≤ 1 cm and asymptomatic are allowed.
* Participants who received a transfusion (platelets, red blood cells) or hematopoetic growth factors within 4 weeks of study treatment.
* Presence of any of the following cardiac criteria/factors:
* Resting QT interval of >470 msec.
* Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG, such as complete left bundle branch block, third degree heart block, or second degree heart block.
* Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death under 40 years of age in first degree relatives, or any concomitant medication known to prolong the QT interval.
* Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required corticosteroid treatment, or any evidence of clinically active interstitial lung disease.
* Participants with known hypersensitivity to the components or excipients of niraparib or osimertinib.
* Participants may not have received prior treatment with anti-PD1, -PDL1, or -CTLA4 inhibitors.
* Participants with a second, clinically active, malignancy. Participants must not have known history or current diagnosis of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML).
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, myocardial infarction, major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, or psychiatric illness/social situations that would limit compliance with study requirements.
* Participants must not have had any known Grade 3 or 4 anemia, neutropenia or thrombocytopenia due to prior chemotherapy that persisted > 4 weeks and was related to the most recent treatment.
* Participants must not have current evidence of any condition, therapy, or laboratory abnormality (including active or uncontrolled myelosuppression [ie, anemia, leukopenia, neutropenia, thrombocytopenia]) that might confound the results of the study or interfere with the patient's participation for the full duration of the study treatment or that makes it not in the best interest of the patient to participate in the opinion of the investigator or sponsor.
* Patients must not have known, active hepatitis B/C.
* Known disorder affecting gastrointestinal absorption.
* Patients must not be pregnant or breastfeeding, or expecting to conceive children, within the projected duration of the study treatment, or for 180 days after the last dose of study treatment.
* Known HIV-positive participants are ineligible because of the potential for pharmacokinetic interactions with Niraparib. In addition, these participants may be at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated, However, HIV testing is not required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-06-06 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose of Niraparib | 2 years

SECONDARY OUTCOMES:
Rate of toxicity of combined niraparib and osimertinib | 2 years
Objective response rate of niraparib | 2 years
Median Progression Free Survival time of Niraparib | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Zofia Piotrowska, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Beth Israel Deaconess, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: BCH - Contact the Technology & Innovation Development Office at www.childrensinnovations.org or email TIDO@childrens.harvard.edu BIDMC - Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu BWH - Contact the Partners Innovations team at http://www.partners.org/innovation DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu MGH - Contact the Partners Innovations team at http://www.partners.org/innovation